CLINICAL TRIAL: NCT01004458
Title: Randomized Clinical Trial of Cognitive Behavioral Therapy in Women With the Fibromyalgia Disorder
Brief Title: Cognitive Behavioral Therapy Trial in Fibromyalgia
Acronym: (FIBCOG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala County Council, Sweden (Other Government); National Social Insurance Board, Sweden (Unknown); The Swedish Society of Medicine (Other); Reumatikerförbundet (Unknown)
Responsible Party: Bo Karlsson, MD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCC2000
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; cognitive behavioral therapy; women; pain; stress; type A behavior
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early treatment group (Active Comparator): The experimental group receiving CBT
  Interventions: Behavioral: Cognitive behavioral therapy
- Waiting list group (No Intervention): The waiting list group served as referents during the trial
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — The treatment, adopted to reduce hostility and stress behavior, was given during group sessions once a week during six months with two follow-up occasions during the next six months
  Arms: Early treatment group
Other: Waiting list — The group served as referents during the trial and received no intervention other than measurements at the same points in time as the intervention group
  Arms: Waiting list group

SUMMARY:
Previous studies have shown that the disorder fibromyalgia often is preceded by long-term stress. Moreover, an association has been shown between stress, pain and co-morbidity in these patients. Cognitive behavioral therapy (CBT) has been shown effective in reducing stress, anxiety and pain in rheumatoid arthritis and fibromyalgia. The purpose of the present trial was to assess whether CBT may reduce pain and other symptoms and increase well-being and general function, affect biological markers for pain and long-term stress, to a larger extent than treatment "as usual".

Forty eight women with verified fibromyalgia were randomly allocated to an early treatment group or a waiting list group. The early treatment group received CBT group treatment during six months. Measurements of outcome and potential outcome affecting variables were made at baseline, after six months and one year after baseline. The waiting list group received the same CBT treatment as the early treatment group after six months on the waiting list.

The design is thus a traditional "waiting list design", allowing a two parallel group comparison during the first six months and a "before-after" analysis in both groups when the treatment was concluded.

DETAILED DESCRIPTION:
Long-lasting pain is a common cause for disability. In several studies 30-40% of the adult general population suffer from pain. In this group of subjects the fibromyalgia syndrome (FMS) is common,. This is a well defined disorder with generalized pain, well defined tenderpoints according to the American Collage of Rheumatology (ACR) criteria, and a number of other associated symptoms. About 5-10% of the general female population suffers from fibromyalgia. The disorder is infrequent among men.

The etiology of the condition is unknown. However, a multi-factorial origin is postulated, where some form of stress is a contributing factor. Also neuro-endocrine disturbances have been observed. Cognitive behavioral therapy CBT) is an evidence based efficient treatment method in depression and panic disorder. In open studies it has proved to be an effective stress and pain reducer.

The purpose of the trial was to evaluate the effect of CBT in a group of female FMS patients regarding pain, stress, and well-being (outcome). A purpose was also to study mediating factors, such as biological markers for stress and pain, and psycho-social factors.

The study population consisted of 48 women, 27-62 years of age, living in Östhammar municipality, central Sweden, with a verified FMS according to the 1992 ACR criteria, and no other serious disorder. The were recruited by advertising in the local printed press and meetings with the local rheumatology patient association.

54 subjects were screened for participation. A physical examination was performed, a medical history was taken, blood samples and saliva specimens for biological markers regarding metabolic status, pain and stress were taken, and a questionnaire was filled out. 48 women fulfilled the inclusion criteria and gave informed consent to participation. A randomized block design was used by which the women were randomly allocated to two groups, an early treatment group and a waiting list group.

The early treatment group was subdivided into four treatment groups with six participants in each. The CBT treatment was given by certified therapists and supervised by the chief therapist, an experienced psychologist. Each group had the same therapist throughout the trial. The therapy was given as group sessions once a week for 20 weeks. When the therapy was completed the outcome variables were measured by means of questionnaire, and the same blood and saliva specimens as at baseline were taken. During the next six months two booster CBT sessions were performed. One year after baseline a final follow-up evaluation was made.

The waiting list group served as reference (or control) group to the early treatment group during the first six months from baseline. No CBT therapy was given, but otherwise exactly the same procedure was followed. When the control period was over the waiting list group got their CBT treatment and evaluations following the same protocol as the early treatment group.

The outcome evaluation are based on a number of questionnaire instruments, such as the Multidimensional Pain Inventory (MPI), the Type A behavior instrument (Everyday stress), The Maastricht Questionnaire ("Vital exhaustion"), and the self administered Montgomery Åsberg Depression Rating Scale (MADRS-S) instrument. The blood sampling aimed at analyzing the neuro-peptides substance P, Met-Enkephalin-Arginine-Phenylalanine (MEAP), beta-endorphin, and neuro-peptide Y, in addition to estrogen, testosterone, prolactin and dehydroepiandrosterone (DHEA). The saliva specimens were intended to measure diurnal variation of cortisol. To standardize the hormonal level all evaluations were done in ovulation phase of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia according to the American College of Rheumatology criteria
* Women
* Age 18-65
* Living in Östhammar municipality, Sweden
* Swedish speaking

Exclusion Criteria:

* severe mental disease
* drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-01; Primary Completion 2003-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Multidimensional Pain Inventory (MPI) score | At baseline and at 6 and 12 months after baseline

SECONDARY OUTCOMES:
Type A behavior measures | At baseline and at 6 and 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bo Karlsson, MD, Principal Investigator — Uppsala University
Locations (1):
- Dept of Public Health and Caring Sciences, Family Medicin and Clinical Epidemiology Section, Uppsala, Sweden

REFERENCES:
- [Derived] Karlsson B, Nyberg F, Svardsudd K, Burell G, Bjorkegren K, Kristiansson P. Neuropeptide Y and measures of stress in a longitudinal study of women with the fibromyalgia syndrome. Scand J Pain. 2022 Jun 21;23(1):59-65. doi: 10.1515/sjpain-2022-0016. Print 2023 Jan 27. PMID 35728621
- See also: Link to department website where the study is briefly described — http://www.pubcare.uu.se